CLINICAL TRIAL: NCT01283516
Title: A Phase I, Multi-center, Open Label Dose Escalation Study of LDK378, Administered Orally in Adult Patients With Tumors Characterized by Genetic Abnormalities in Anaplastic Lymphoma Kinase (ALK)
Brief Title: A Dose Escalation/Expansion Study of LDK378 in Patients With Tumors Characterized by Genetic Abnormalities in Anaplastic Lymphoma Kinase
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLDK378X2101; 2010-019827-70 (EudraCT Number)
Record Dates: First submitted 2011-01-24; First posted 2011-01-26 (Estimated); Results first posted 2014-08-11 (Estimated); Last update posted 2019-03-15 (Actual); Status verified 2018-11

CONDITIONS: Tumors Characterized by Genetic Abnormalities of ALK
Keywords: ALK inhibitor,; NSCLC,; LDK378,; ceritinib,; genetic abnormalities
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ceritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LDK378 750 mg: Arm 1A and Arm 1B (Experimental): NSCLC patients previously treated with an ALK inhibitor
  Interventions: Drug: LDK378
- LDK378 750 mg: Arm 2 (Experimental): NSCLC patients not previously treated with an ALK inhibitor
  Interventions: Drug: LDK378
- LDK378 750 mg: Arm 3 (Experimental): Patients with other tumors that are ALK positive other than NSCLC
  Interventions: Drug: LDK378

INTERVENTIONS:
Drug: LDK378 — LDK378 is a selective and a potent inhibitor of anaplastic lymphoma kinase (ALK) activity, is a capsule and is administered orally.

SUMMARY:
This study assessed the safety and efficacy of LDK378 in adult patients with genetic abnormalities in anaplastic lymphoma kinase (ALK).

ELIGIBILITY:
Inclusion Criteria:

* ECOG Performance Status of ≤ 2 and life expectancy of ≥ 12 weeks.
* Diagnosed with a locally advanced or metastatic malignancy that has progressed despite standard therapy, or for which no effective standard therapy exists. Only patients with tumors characterized by genetic abnormalities in ALK were enrolled.
* For NSCLC, an ALK translocation must be detected by FISH in ≥ 15% of tumor cells.
* In patients with diseases other than NSCLC, ALK translocation is not required and overexpression of ALK protein may be considered indicative of a genetic abnormality in ALK.
* Patients with measurable or non-measurable disease as determined by modified RECIST version 1.0 in dose-escalation phase, and patients with at least one measurable lesion as determined by RECIST 1.0 in expansion phase.

Exclusion Criteria:

* Patients with symptomatic central nervous system (CNS) metastases who were neurologically unstable or required increasing doses of steroids to control their CNS disease were excluded.
* Patients with a prior or current history of a second malignancy, impaired GI function, history of pancreatitis or increased amylase or lipase, known diagnosis of HIV, and clinically significant cardiac disease were excluded.
* Patients treated with chemotherapy or biologic therapy or other investigational agent < 2 weeks prior to starting study drug for compounds with a half-life ≤ 3 days, and < 4 weeks prior to starting study drug for compounds with a prolonged half-life were excluded.
* Further, patients treated with medications that were known to be strong inhibitors or inducers of CYP3A4/5 that could not be discontinued at least a week prior to start of treatment with LDK378 and for the duration of the study were also excluded.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2011-01-24 (Actual); Primary Completion 2016-05-03 (Actual); Study Completion 2016-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (21):
- United States (6):
  - University of Colorado School of Medicine Colorado Univ, Aurora, Colorado
  - Massachusetts General Hospital Mass General, Boston, Massachusetts
  - Memorial Sloan Kettering MSK, New York, New York
  - Fox Chase Cancer Center Fox Chase Cancer (2), Philadelphia, Pennsylvania
  - University of Utah / Huntsman Cancer Institute Huntsman, Salt Lake City, Utah
  - Seattle Cancer Care Alliance, Seattle, Washington
- Novartis Investigative Site, Melbourne, Victoria, Australia
- Novartis Investigative Site, Leuven, Belgium
- Novartis Investigative Site, Toronto, Ontario, Canada
- Germany (4):
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Ulm
- Italy (2):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
- Novartis Investigative Site, Amsterdam, Netherlands
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Seoul, Korea, South Korea
- Novartis Investigative Site, Barcelona, Catalonia, Spain
- United Kingdom (2):
  - Novartis Investigative Site, Glasgow, Scotland
  - Novartis Investigative Site, Leicester

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tan DS, Thomas M, Kim DW, Szpakowski S, Urban P, Mehra R, Chow LQM, Sharma S, Solomon BJ, Felip E, Camidge DR, Vansteenkiste J, Petruzzelli L, Pantano S, Shaw AT. Genetic landscape of patients with ALK-rearranged non-small-cell lung cancer (NSCLC) and response to ceritinib in ASCEND-1 study. Lung Cancer. 2022 Jan;163:7-13. doi: 10.1016/j.lungcan.2021.11.007. Epub 2021 Nov 20. PMID 34890832
- [Derived] Kim DW, Mehra R, Tan DSW, Felip E, Chow LQM, Camidge DR, Vansteenkiste J, Sharma S, De Pas T, Riely GJ, Solomon BJ, Wolf J, Thomas M, Schuler M, Liu G, Santoro A, Sutradhar S, Li S, Szczudlo T, Yovine A, Shaw AT. Activity and safety of ceritinib in patients with ALK-rearranged non-small-cell lung cancer (ASCEND-1): updated results from the multicentre, open-label, phase 1 trial. Lancet Oncol. 2016 Apr;17(4):452-463. doi: 10.1016/S1470-2045(15)00614-2. Epub 2016 Mar 11. PMID 26973324
- [Derived] Richly H, Kim TM, Schuler M, Kim DW, Harrison SJ, Shaw AT, Boral AL, Yovine A, Solomon B. Ceritinib in patients with advanced anaplastic lymphoma kinase-rearranged anaplastic large-cell lymphoma. Blood. 2015 Sep 3;126(10):1257-8. doi: 10.1182/blood-2014-12-617779. No abstract available. PMID 26337354
- [Derived] Shaw AT, Kim DW, Mehra R, Tan DS, Felip E, Chow LQ, Camidge DR, Vansteenkiste J, Sharma S, De Pas T, Riely GJ, Solomon BJ, Wolf J, Thomas M, Schuler M, Liu G, Santoro A, Lau YY, Goldwasser M, Boral AL, Engelman JA. Ceritinib in ALK-rearranged non-small-cell lung cancer. N Engl J Med. 2014 Mar 27;370(13):1189-97. doi: 10.1056/NEJMoa1311107. PMID 24670165
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/26272586

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was considered completed when all patients discontinued ceritinib treatment, & all required follow-up was completed or patient died, was lost to follow-up or withdrew their consent to further participate in study or last patient on treatment was enrolled to a separate protocol to continue receiving ceritinib treatment, whichever came first.
Pre-assignment Details: A total of 304 patients were treated with LDK378 in the study, including 59 patients from the dose-escalation phase (including 10 patients at 750 mg) and 245 patients from the expansion phase treated at LDK378 750 mg.
Groups:
- LDK378 50 mg: Participants receiving 50 mg of LDK378
- LDK378 100 mg: Participants receiving 100 mg of LDK378
- LDK378 200 mg: Participants receiving 200 mg of LDK378
- LDK378 300 mg: Participants receiving 300 mg of LDK378
- LDK378 400 mg: Participants receiving 400 mg of LDK378
- LDK378 500 mg: Participants receiving 500 mg of LDK378
- LDK378 600 mg: Participants receiving 600 mg of LDK378
- LDK378 700 mg: Participants receiving 700 mg of LDK378
- LDK378 750 mg: Participants receiving 750 mg of LDK378.
Period: Overall Study
Arm/Group | LDK378 50 mg | LDK378 100 mg | LDK378 200 mg | LDK378 300 mg | LDK378 400 mg | LDK378 500 mg | LDK378 600 mg | LDK378 700 mg | LDK378 750 mg
Started | 2 (Started = Full Analysis Set and Safety Set) | 2 | 3 | 3 | 14 | 10 | 10 | 5 | 255
Non-Small Cell Lung Cancer (NSCLC) | 2 | 1 | 2 | 3 | 12 | 10 | 9 | 5 | 246
Dose-Determining Set (DDS) | 2 | 1 | 3 | 3 | 14 | 8 | 10 | 5 | 8
Non-NSCLC | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 9 (Small number of patients at 750 mg - non-NSCLC, assessment limited, not included in efficacy tables)
Completed | 0 (Completed - see explanation in Recruitment Details.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 2 | 3 | 3 | 14 | 10 | 10 | 5 | 255
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 28
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 12
Not completed — Disease Progression | 2 | 2 | 3 | 3 | 13 | 8 | 6 | 3 | 139
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 36
Not completed — Administrative problems | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 39
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) consisted of all patients (including NSCLC and non-NSCLC) who received at least one dose of LDK378. Patients were classified according to the intended treatment dose group.
Groups:
- Total: Total of all reporting groups
Arm/Group | LDK378 50 mg | LDK378 100 mg | LDK378 200 mg | LDK378 300 mg | LDK378 400 mg | LDK378 500 mg | LDK378 600 mg | LDK378 700 mg | LDK378 750 mg | Total
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 14 | 10 | 10 | 5 | 255 | 304
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.5 (23.33) | 30.5 (12.02) | 53.7 (10.69) | 58.7 (5.03) | 48.7 (15.62) | 55.0 (15.99) | 54.6 (13.22) | 56.4 (4.67) | 51.9 (12.08) | 52.0 (12.41)
Age, Customized [Number; unit: Participants]
  <65 years | 2 | 2 | 2 | 3 | 12 | 7 | 7 | 5 | 215 | 255
  >=65 years | 0 | 0 | 1 | 0 | 2 | 3 | 3 | 0 | 40 | 49
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 3 | 2 | 10 | 6 | 7 | 4 | 136 | 170
  Male | 1 | 1 | 0 | 1 | 4 | 4 | 3 | 1 | 119 | 134
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 1 | 26 | 32
  Chinese | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 17 | 19
  Indian (Indian subcontinent) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
  Mixed Ethnicity | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 3
  Other | 2 | 2 | 2 | 3 | 12 | 8 | 6 | 4 | 205 | 244
Predominant Race [Number; unit: Participants]
  Caucasian | 2 | 2 | 2 | 2 | 12 | 8 | 8 | 3 | 160 | 199
  Black | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4
  Asian | 0 | 0 | 0 | 1 | 2 | 2 | 2 | 1 | 87 | 95
  Native American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Pacific Islander | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 4
Weight [Mean (Standard Deviation); unit: Kilograms (kg)] | 60.8 (19.80) | 67.8 (5.94) | 69.2 (17.20) | 54.1 (9.70) | 69.2 (15.91) | 72.2 (18.74) | 63.8 (13.23) | 61.6 (16.05) | 69.2 (15.64) | 68.8 (15.61)
Height [Mean (Standard Deviation); unit: centimenters (cm)] — Population: Full Analysis Set (FAS) consisted of all patients (including NSCLC and non-NSCLC) who received at least one dose of LDK378. Height was not collected for 1 patient each in the 700 mg arm and the 750 mg arm.
  centimenters (cm)
    number analyzed (Participants) | 2 | 2 | 3 | 3 | 14 | 10 | 10 | 4 | 254 | 302
    (all) | 169.0 (7.07) | 178.0 (14.14) | 161.3 (3.04) | 164.6 (5.82) | 169.9 (9.35) | 166.4 (12.24) | 165.1 (8.67) | 163.6 (5.05) | 167.5 (9.87) | 167.5 (9.78)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: Full Analysis Set (FAS) consisted of all patients (including NSCLC and non-NSCLC) who received at least one dose of LDK378. Body Mass Index was not collected for 1 patient each in the 700 mg arm and the 750 mg arm.
  kg/m^2
    number analyzed (Participants) | 2 | 2 | 3 | 3 | 14 | 10 | 10 | 4 | 254 | 302
    (all) | 21.1 (5.16) | 21.8 (5.30) | 26.5 (5.69) | 20.2 (5.08) | 24.0 (5.38) | 25.9 (5.41) | 23.1 (2.78) | 24.3 (6.06) | 24.5 (4.40) | 24.4 (4.48)
WHO/ECOG Performance status [Number; unit: Participants] — The ECOG performance status is a scale used to assess how a patient's disease is progressing, assess how the disease affects the daily living abilities of the patient, and determine appropriate treatment and prognosis.
  Participants
    0:Fully active,in line with pre-disease activities | 1 | 1 | 1 | 0 | 3 | 2 | 2 | 1 | 65 | 76
    1: Able to carry out light work | 1 | 1 | 2 | 3 | 8 | 7 | 7 | 3 | 161 | 193
    2:Capable of self-care up & about >50% of the time | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 1 | 28 | 34
    3: Limited self-care, confined to bed/chair >50% | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Smoking History [Number; unit: Participants]
  Never Smoked | 2 | 1 | 1 | 2 | 9 | 7 | 8 | 3 | 159 | 192
  Ex-Smoker | 0 | 1 | 2 | 1 | 5 | 3 | 2 | 2 | 88 | 104
  Current Smoker | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: The maximum tolerated dose (MTD) was defined as the highest dose for a given schedule that was expected to cause DLTs in no more than 33% of patients during the first cycle of treatment. A patient with multiple occurrences of a DLT under one treatment is counted only once in the AE category for that treatment. MTD was determined at 750mg.
Time Frame: 33 months
Population: Dose-determining Set (DDS) consists of all patients (NSCLC and non-NSCLC) from the safety set who either meet the minimum exposure criterion and have sufficient safety evaluations or have experienced a dose limiting toxicity (DLT) during Cycle 1 (including the PK run-in period). This constitutes all evaluable patients for the determination of MTD.
Measure: Number; unit: Participants
Arm/Group | LDK378 50 mg | LDK378 100 mg | LDK378 200 mg | LDK378 300 mg | LDK378 400 mg | LDK378 500 mg | LDK378 600 mg | LDK378 700 mg | LDK378 750 mg
Number analyzed (Participants) | 2 | 1 | 3 | 3 | 14 | 8 | 10 | 5 | 8
Participants
  Diarrhea | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Vomiting | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Alanine Aminotransferase Increased | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Transaminases Increased | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Dehydration | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Hypophosphataemia | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

2. Secondary Outcome: Overall Response Rate (ORR) Based on Investigator Assessment
Description: Overall response rate (ORR) was defined as the percentage of participants with a best overall complete response (CR) or partial response (PR) per RECIST 1.0. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI. Both CR and PR had to be confirmed by repeat assessments performed no less than 4 weeks after the criteria for response were first met. CR was the disappearance of all target lesions. PR was at least a 30% decrease in the sum of the longest diameter of all target lesions, taking as reference the baseline sum of the longest diameters. Both CR and PR had to be confirmed by repeat assessments performed no less than 4 weeks after the criteria for response were first met. CR = at least two determinations of CR, at least 4 weeks apart before progression. PR = at least two determinations of PR or better at least 4 weeks apart before progression (and not qualifying for a CR).
Time Frame: 275 weeks
Population: Full analysis set (FAS) - NSCLC: Subset of Full Analysis Set including ALK-positive NSCLC patients who received at least one dose of LDK378 in the 750 mg dose group.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- NSCLC With Prior ALKi (Arms 1A + 1B): Patients with ALK-translocated NSCLC who were previously treated with an ALK inhibitor.
- NSCLC ALKi Naive (Arm 2): Patients with ALK-translocated NSCLC not previously treated with an ALK inhibitor.
- All NSCLC: all NSCLC patients.
Arm/Group | NSCLC With Prior ALKi (Arms 1A + 1B) | NSCLC ALKi Naive (Arm 2) | All NSCLC
Number analyzed (Participants) | 163 | 83 | 246
Percentage of Participants | 56.4 [48.5 to 64.2] | 73.5 [62.7 to 82.6] | 62.2 [55.8 to 68.3]

3. Secondary Outcome: Overall Response Rate Based on Blinded Independent Review Committee (BIRC) Assessment
Description: Overall response rate (ORR) was defined as the percentage of participants with a best overall complete response (CR) or partial response (PR) per RECIST 1.0. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI, CR was the disappearance of all target lesions. PR was at least a 30% decrease in the sum of the longest diameter of all target lesions, taking as reference the baseline sum of the longest diameters. Both CR and PR had to be confirmed by repeat assessments performed no less than 4 weeks after the criteria for response were first met. CR = at least two determinations of CR, at least 4 weeks apart before progression. PR = at least two determinations of PR or better at least 4 weeks apart before progression (and not qualifying for a CR).
Time Frame: 275 weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- All NCSLC: all NSCLC patients.
Arm/Group | NSCLC With Prior ALKi (Arms 1A + 1B) | NSCLC ALKi Naive (Arm 2) | All NCSLC
Number analyzed (Participants) | 163 | 83 | 246
Percentage of participants | 49.1 [41.2 to 57.0] | 65.1 [53.8 to 75.2] | 54.5 [48.0 to 60.8]

4. Secondary Outcome: Duration of Response (DOR) Based on Investigator Assessment
Description: Duration of response (DOR) was defined as the time from first documented response (partial response (PR) or complete response (CR)) to the date of first documented disease progression (PD) or death due to any cause, among patients with a confirmed PR or CR per RECIST 1.0.
Time Frame: 275 weeks
Population: Full analysis set (FAS) - NSCLC: Subset of Full Analysis Set including ALK-positive NSCLC patients who received at least one dose of LDK378 in the 750 mg dose group and had a confirmed overall complete response or partial response after initiation of LDK378.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NSCLC With Prior ALKi (Arms 1A + 1B) | NSCLC ALKi Naive (Arm 2) | All NSCLC
Number analyzed (Participants) | 92 | 61 | 153
months | 8.25 [6.80 to 9.69] | 14.19 [11.27 to 22.11] | 10.12 [8.31 to 11.63]

5. Secondary Outcome: Duration of Response (DOR) Based on BIRC
Description: as for outcome 4
Time Frame: 275 weeks
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NSCLC With Prior ALKi (Arms 1A + 1B) | NSCLC ALKi Naive (Arm 2) | All NSCLC
Number analyzed (Participants) | 80 | 54 | 134
months | 8.31 [5.98 to 12.42] | 21.75 [14.06 to 31.11] | 12.45 [8.77 to 16.56]

6. Secondary Outcome: Progression-free Survival Based on Investigator Assessment
Description: Progression-free survival (PFS) was defined as the time from the start date of study drug to the date of the first radiologically documented progressive disease (PD) per RECIST 1.0. or death due to any cause.
Time Frame: 275 weeks
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NSCLC With Prior ALKi (Arms 1A + 1B) | NSCLC ALKi Naive (Arm 2) | All NSCLC
Number analyzed (Participants) | 163 | 83 | 246
months | 6.93 [5.55 to 8.48] | 15.21 [12.12 to 19.48] | 8.74 [6.93 to 10.97]

7. Secondary Outcome: Progression-free Survival Based on BIRC Assessment
Description: as for outcome 6
Time Frame: 275 weeks
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NSCLC With Prior ALKi (Arms 1A + 1B) | NSCLC ALKi Naive (Arm 2) | ALL NSCLC
Number analyzed (Participants) | 163 | 83 | 246
months | 6.97 [5.55 to 8.57] | 19.32 [11.99 to 29.01] | 9.53 [7.00 to 11.50]

8. Secondary Outcome: Primary Pharmacokinetics (PK) Parameter: AUC0-last
Description: The AUC from time zero to the last quantifiable concentration point (Tlast). Blood samples for PK analysis of LDK378 were collected during the study from patients receiving LDK378.
Time Frame: PK run-in of Dose Escalation phase
Population: Pharmacokinetic Analysis Set (PAS) consisted of all patients (including NSCLC and non-NSCLC) who received at least 1 dose of LDK378 & had at least 1 evaluable PK sample
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | LDK378 50 mg | LDK378 100 mg | LDK378 200 mg | LDK378 300 mg | LDK378 400 mg | LDK378 500 mg | LDK378 600 mg | LDK378 700 mg | LDK378 750 mg
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 14 | 10 | 10 | 5 | 252
ng*h/mL | 366 (NA) — N/A = not estimable | 938 (24.3) | 1460 (62.9) | 7470 (46.5) | 4070 (81.8) | 5140 (141.7) | 8180 (57.4) | 9210 (111.7) | 7870 (127.3)

9. Secondary Outcome: Primary Pharmacokinetics (PK) Parameter: AUC0-24h
Description: Blood samples for PK analysis of LDK378 were collected during the study from patients receiving LDK378. AUC0 - 24 is the AUC calculated to 24 hour. Cycle 1 Day 1 = C1D1; Cycle 1 Day 8 = C1D8; Cycle 2 Day 1 = C2D1. However, there was no PK sampling during C1D1 and C2D1 except for 750 mg dose to compute PK parameter AUC0-24.
Time Frame: PK run-in of dose escalation phase, Cycle 1 Day 8 of dose escalation phase, Cycle 1, Day 1 of dose escalation phase, Cycle 2 Day 1 of dose escalation & dose expansion phases
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | LDK378 50 mg | LDK378 100 mg | LDK378 200 mg | LDK378 300 mg | LDK378 400 mg | LDK378 500 mg | LDK378 600 mg | LDK378 700 mg | LDK378 750 mg
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 14 | 10 | 10 | 5 | 252
ng*h/mL
  PK Run-in dose escalation phase: number analyzed (Participants) | 1 | 2 | 2 | 3 | 12 | 8 | 9 | 4 | 10
  PK Run-in dose escalation phase | 226 (NA) — N/A = not estimable | 467 (10.7) | 703 (55.6) | 3440 (44.7) | 1920 (78.0) | 2350 (87.9) | 3590 (53.4) | 3450 (137.9) | 3390 (121.4)
  C1D8: dose escalation phase: number analyzed (Participants) | 2 | 2 | 3 | 2 | 9 | 9 | 7 | 2 | 8
  C1D8: dose escalation phase | 435 (42.1) | 1520 (41.1) | 4150 (32.2) | 7660 (402.8) | 7680 (77.4) | 12300 (37.4) | 14700 (71.7) | 35200 (0.800) | 13900 (74.8)
  C1D1 dose escalation phase for 750mg: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 73
  C1D1 dose escalation phase for 750mg |  |  |  |  |  |  |  |  | 3340 (111.9)
  C2D1 dose escalation & expansion phases: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 23
  C2D1 dose escalation & expansion phases | 376 (NA) — N/A = not estimable | 894 (NA) — N/A = not estimable |  |  |  |  |  |  | 22600 (37.1)

10. Secondary Outcome: Primary Pharmacokinetics (PK) Parameter: Tmax
Description: Tmax is the time to reach Cmax. Blood samples for PK analysis of LDK378 were collected during the study from patients receiving LDK378. Blood samples for PK analysis of LDK378 were collected during the study from patients receiving LDK378. Cycle 1 Day 1 = C1D1; Cycle 1 Day 8 = C1D8; Cycle 2 Day 1 = C2D1. However, there was no PK sampling during C1D1 and C2D1 except for 750 mg dose to compute PK parameter Tmax.
Time Frame: as for outcome 9
Population: as for outcome 8
Measure: Median (Full Range); unit: hour
Arm/Group | LDK378 50 mg | LDK378 100 mg | LDK378 200 mg | LDK378 300 mg | LDK378 400 mg | LDK378 500 mg | LDK378 600 mg | LDK378 700 mg | LDK378 750 mg
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 14 | 10 | 10 | 5 | 252
hour
  PK run-in dose escalation phase: number analyzed (Participants) | 1 | 2 | 2 | 3 | 12 | 8 | 9 | 4 | 10
  PK run-in dose escalation phase | 5.95 [5.95 to 5.95] | 15.0 [6.00 to 24.0] | 5.08 [4.17 to 6.00] | 4.00 [4.00 to 5.95] | 4.99 [2.97 to 6.73] | 3.98 [3.00 to 23.5] | 6.00 [3.00 to 24.1] | 6.00 [4.00 to 25.0] | 6.02 [3.95 to 23.8]
  C1D8 dose escalation phase: number analyzed (Participants) | 2 | 2 | 3 | 3 | 13 | 9 | 9 | 5 | 8
  C1D8 dose escalation phase | 2.46 [2.00 to 2.92] | 3.49 [3.00 to 3.98] | 3.00 [2.98 to 7.95] | 4.00 [3.00 to 7.18] | 6.08 [2.98 to 24.0] | 3.95 [1.93 to 6.00] | 4.00 [0.00 to 23.6] | 5.97 [2.00 to 24.0] | 5.03 [3.00 to 7.95]
  C1D1 dose escalation phase for 750mg: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 208
  C1D1 dose escalation phase for 750mg |  |  |  |  |  |  |  |  | 6.00 [1.13 to 24.0]
  C2D1 dose escalation & dose expansion phases: number analyzed (Participants) | 2 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 133
  C2D1 dose escalation & dose expansion phases | 5.00 [4.00 to 6.00] | 2.08 [2.08 to 2.08] | 8.00 [4.00 to 23.9] |  |  |  |  |  | 6.00 [0.00 to 22.6]

11. Secondary Outcome: Primary Pharmacokinetics (PK) Parameter: Cmax
Description: Cmax is the maximum observed concentration. Blood samples for PK analysis of LDK378 were collected during the study from patients receiving LDK378. However, there was no PK sampling during C1D1 and C2D1 except for 750 mg dose to compute PK parameter Cmax.
Time Frame: PK run-in of dose escalation phase, Cycle 1 Day 8 of dose escalation phase, Cycle 1, Day 1 of dose escalation ion phase, Cycle 2 Day 1 of dose escalation & expansion phases
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | LDK378 50 mg | LDK378 100 mg | LDK378 200 mg | LDK378 300 mg | LDK378 400 mg | LDK378 500 mg | LDK378 600 mg | LDK378 700 mg | LDK378 750 mg
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 14 | 10 | 10 | 5 | 252
ng/mL
  PK Run-in dose escalation phase: number analyzed (Participants) | 1 | 2 | 2 | 3 | 12 | 8 | 9 | 4 | 10
  PK Run-in dose escalation phase | 13.1 (NA) — N/A = not estimable | 29.3 (10.1) | 40.2 (88.5) | 198 (41.5) | 120 (80.9) | 153 (86.5) | 212 (59.7) | 206 (145.6) | 186 (126.9)
  C1D8 dose escalation phase: number analyzed (Participants) | 2 | 2 | 3 | 3 | 13 | 9 | 9 | 5 | 8
  C1D8 dose escalation phase | 25.1 (37.5) | 76.7 (20.9) | 212 (18.0) | 381 (167.5) | 419 (69.7) | 641 (40.0) | 688 (68.3) | 1140 (37.7) | 674 (76.2)
  C1D1 dose escalation phase for 750mg: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 208
  C1D1 dose escalation phase for 750mg |  |  |  |  |  |  |  |  | 203 (100.9)
  C2D1 dose escalation & dose expansion phases: number analyzed (Participants) | 2 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 133
  C2D1 dose escalation & dose expansion phases | 21.9 (9.4) | 53.5 (NA) — N/A = not estimable | 229 (120.7) |  |  |  |  |  | 1010 (44.8)

12. Secondary Outcome: Secondary Pharmacokinetics (PK) Parameter: T1/2
Description: T1/2 is the elimination half-life associated with the terminal slope (λz) of a semi logarithmic concentration-time curve (time). Blood samples for PK analysis of LDK378 were collected during the study from patients receiving LDK378. Blood samples for PK analysis of LDK378 were collected during the study from patients receiving LDK378.
Time Frame: PK Run-in dose escalation phase
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | LDK378 50 mg | LDK378 100 mg | LDK378 200 mg | LDK378 300 mg | LDK378 400 mg | LDK378 500 mg | LDK378 600 mg | LDK378 700 mg | LDK378 750 mg
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 10 | 7 | 6 | 3 | 9
hour | 19.5 (NA) — N/A = not estimable | 19.4 (NA) — N/A = not estimable | 33.2 (NA) — N/A = not estimable | 30.1 (10.0) | 30.7 (39.1) | 31.1 (11.1) | 37.6 (24.6) | 38.9 (98.4) | 40.6 (34.7)

13. Secondary Outcome: Secondary Pharmacokinetics (PK) Parameter: CL/F
Description: CL/F is the apparent total body clearance of drug from the plasma
Time Frame: PK Run-in dose escalation phase
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litres/hour
Arm/Group | LDK378 50 mg | LDK378 100 mg | LDK378 200 mg | LDK378 300 mg | LDK378 400 mg | LDK378 500 mg | LDK378 600 mg | LDK378 700 mg | LDK378 750 mg
Number analyzed (Participants) | 1 | 1 | 1 | 2 | 5 | 3 | 2 | 2 | 3
Litres/hour | 126 (NA) — N/A = not estimable | 116 (NA) — N/A = not estimable | 77.5 (NA) — N/A = not estimable | 44.5 (36.8) | 95.9 (58.6) | 147.0 (170.3) | 46.3 (9.6) | 66.6 (35.8) | 88.5 (162.5)

14. Secondary Outcome: Secondary Pharmacokinetics (PK) Parameter: Vz/F
Description: Vz/F is the apparent volume of distribution during terminal phase (associated with Lambda_z)
Time Frame: PK Run-in dose escalation phase
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litre
Arm/Group | LDK378 50 mg | LDK378 100 mg | LDK378 200 mg | LDK378 300 mg | LDK378 400 mg | LDK378 500 mg | LDK378 600 mg | LDK378 700 mg | LDK378 750 mg
Number analyzed (Participants) | 1 | 1 | 1 | 2 | 5 | 3 | 2 | 2 | 3
Litre | 3540 (NA) — N/A = not estimable | 3250 (NA) — N/A = not estimable | 3720 (NA) — N/A = not estimable | 1880 (50.7) | 3470 (74.4) | 6230 (218.9) | 1990 (4.3) | 2340 (56.5) | 4230 (164.4)

15. Secondary Outcome: Secondary Pharmacokinetics (PK) Parameter: CLss/F
Description: CLss/F is the apparent total body clearance of drug from the plasma. There was no PK sampling during C1D1 and C2D1 except for 750 mg dose to compute PK parameter CLss/F.
Time Frame: Cycle 1 Day 8 of dose escalation phase, Cycle 2 Day 1 of dose escalation & dose expansion phases
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litres/hour
Arm/Group | LDK378 50 mg | LDK378 100 mg | LDK378 200 mg | LDK378 300 mg | LDK378 400 mg | LDK378 500 mg | LDK378 600 mg | LDK378 700 mg | LDK378 750 mg
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 14 | 10 | 10 | 5 | 252
Litres/hour
  C1D8: dose escalation phase: number analyzed (Participants) | 2 | 2 | 3 | 2 | 9 | 9 | 7 | 2 | 8
  C1D8: dose escalation phase | 115 (42.1) | 65.8 (41.1) | 48.2 (32.2) | 39.2 (402.8) | 52.1 (77.4) | 40.7 (37.4) | 40.8 (71.7) | 19.9 (0.8) | 53.9 (74.8)
  C2D1:dose escalation & dose expansion phases: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 23
  C2D1:dose escalation & dose expansion phases | 133 (NA) — N/A = not estimable | 112 (NA) — N/A = not estimable |  |  |  |  |  |  | 33.2 (37.1)

16. Secondary Outcome: Secondary Pharmacokinetics (PK) Parameter: Racc
Description: Racc is the accumulation ratio calculated using AUCtau values obtained from a dosing interval at steady-state divided by AUCtau at day 1 or PK run-in phase. AUCtau is the AUC calculated to the end of the dosing interval, tau. Blood samples for PK analysis of LDK378 were collected during the study from patients receiving LDK378. Blood samples for PK analysis of LDK378 were collected during the study from patients receiving LDK378. However, there was no PK sampling during C1D1 and C2D1 except for 750 mg dose to compute PK parameter Racc.
Time Frame: Cycle 1 Day 8 of dose escalation phase, Cycle 2 Day 1 of dose escalation & dose expansion phases
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: unitless
Arm/Group | LDK378 50 mg | LDK378 100 mg | LDK378 200 mg | LDK378 300 mg | LDK378 400 mg | LDK378 500 mg | LDK378 600 mg | LDK378 700 mg | LDK378 750 mg
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 14 | 10 | 10 | 5 | 252
unitless
  C1D8: dose escalation phase: number analyzed (Participants) | 1 | 2 | 2 | 2 | 7 | 7 | 6 | 2 | 8
  C1D8: dose escalation phase | 2.56 (NA) — N/A = not estimable | 3.25 (53.5) | 6.62 (17.6) | 1.83 (215.9) | 3.80 (124.7) | 6.08 (71.5) | 3.55 (51.7) | 6.84 (89.4) | 4.68 (72.1)
  C2D1: dose escalation & dose expansion phases: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 9
  C2D1: dose escalation & dose expansion phases | 1.67 (NA) — N/A = not estimable | 1.77 (NA) — N/A = not estimable |  |  |  |  |  |  | 6.20 (58.5)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV), at least 30 days following the last dose of study treatment . All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit) up to approximately 5 years.
Groups:
- All Participants: All participants enrolled in the study
Arm/Group | LDK378 50 mg | LDK378 100 mg | LDK378 200 mg | LDK378 300 mg | LDK378 400 mg | LDK378 500 mg | LDK378 600 mg | LDK378 700 mg | LDK378 750 mg | All Participants
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/2 | 1/3 | 1/3 | 7/14 | 4/10 | 7/10 | 3/5 | 145/255 | 169/304
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 3/3 | 3/3 | 14/14 | 10/10 | 10/10 | 5/5 | 254/255 | 303/304
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LDK378 50 mg (N=2) | LDK378 100 mg (N=2) | LDK378 200 mg (N=3) | LDK378 300 mg (N=3) | LDK378 400 mg (N=14) | LDK378 500 mg (N=10) | LDK378 600 mg (N=10) | LDK378 700 mg (N=5) | LDK378 750 mg (N=255) | All Participants (N=304)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Angina Pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 3
Cardiac Failure Congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cardiac Tamponade (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Cardio-Respiratory Arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pericardial Effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 6 | 7
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5
Stress Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Supraventricular Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Atrial Septal Defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hearing Impaired (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Diabetic Retinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Gastric Ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Gastritis Haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Intestinal Perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Intra-Abdominal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 3 | 6
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Drug Withdrawal Syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Gait Disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
General Physical Health Deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
Multi-Organ Failure (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4
Bile Duct Obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Drug-Induced Liver Injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Gallbladder Fistula (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Gallbladder Oedema (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Gallbladder Perforation (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hepatitis Cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Appendicitis Perforated (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Bacterial Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cranial Nerve Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Empyema (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Ludwig Angina (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Lung Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Neutropenic Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Oral Candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 19 | 20
Pneumonia Bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Pulmonary Tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Septic Shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Compression Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Eye Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Facial Bones Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 5 | 6
Amylase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 4
Blood Creatinine Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Blood Urea Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Ejection Fraction Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Lipase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Oxygen Saturation Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Platelet Count Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Transaminases Increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 5
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Fracture Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Tendon Disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Malignant Neoplasm Of Thorax (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Malignant Pleural Effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Metastases To Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Metastases To Meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Brain Oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Cauda Equina Syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Central Nervous System Necrosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cognitive Disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Depressed Level Of Consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Generalised Tonic-Clonic Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Haemorrhage Intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Loss Of Consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Nervous System Disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Paraplegia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 16 | 18
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Speech Disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Spinal Cord Compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Toxic Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Confusional State (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Mental Disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Mental Status Changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Azotaemia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Calculus Ureteric (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Renal Failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pelvic Pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Asthma-Chronic Obstructive Pulmonary Disease Overlap Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 15 | 16
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Obstructive Airways Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 9
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 5
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 4
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 6 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LDK378 50 mg (N=2) | LDK378 100 mg (N=2) | LDK378 200 mg (N=3) | LDK378 300 mg (N=3) | LDK378 400 mg (N=14) | LDK378 500 mg (N=10) | LDK378 600 mg (N=10) | LDK378 700 mg (N=5) | LDK378 750 mg (N=255) | All Participants (N=304)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 2 | 2 | 3 | 0 | 32 | 40
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 3
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 5 | 6
Sinus Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 5
Sinus Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 3
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 6 | 7
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 7 | 8
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 7 | 8
Blepharospasm (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 5
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 3
Eyelid Ptosis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Photopsia (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 2 | 5
Visual Impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 17
Vitreous Floaters (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 3
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 18 | 19
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 9 | 13
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 3 | 2 | 1 | 102 | 111
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 4
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 64 | 68
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 3 | 3 | 4 | 2 | 90 | 103
Dental Caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 5
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 9 | 7 | 8 | 4 | 221 | 252
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 4 | 1 | 35 | 43
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 7 | 10
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 11 | 12
Gastrointestinal Disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Gastrointestinal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 20 | 22
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 5
Melaena (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Mouth Swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 2 | 2 | 10 | 9 | 10 | 5 | 215 | 254
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 17 | 18
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 5
Vomiting (Gastrointestinal disorders) | 0 | 1 | 3 | 1 | 8 | 5 | 8 | 4 | 159 | 189
Asthenia (General disorders) | 0 | 1 | 1 | 1 | 2 | 1 | 3 | 3 | 58 | 70
Axillary Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest Discomfort (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 23 | 26
Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 18 | 19
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 14 | 15
Facial Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 3
Fatigue (General disorders) | 1 | 1 | 1 | 0 | 5 | 4 | 8 | 1 | 111 | 132
Gait Disturbance (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 10 | 11
Hunger (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Influenza Like Illness (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 6 | 8
Local Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 28 | 30
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 4 | 6
Oedema Peripheral (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 32 | 35
Pain (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 18 | 21
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 46 | 50
Seasonal Allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 6 | 7
Bacterial Disease Carrier (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 7 | 9
Clostridium Difficile Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 5
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Herpes Dermatitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 20 | 22
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 23 | 26
Oral Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 13 | 14
Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 6 | 8
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Tooth Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 3
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 3 | 2 | 1 | 1 | 32 | 40
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 18 | 21
Vaginal Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vulvovaginal Candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Burns First Degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 8 | 10
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 3
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tendon Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 1 | 0 | 2 | 3 | 3 | 4 | 122 | 135
Amylase Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 0 | 23 | 28
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 1 | 0 | 3 | 2 | 3 | 3 | 91 | 103
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 48 | 52
Blood Creatinine Increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 47 | 49
Blood Lactate Dehydrogenase Increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 7
Blood Magnesium Decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
C-Reactive Protein Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 10 | 11
Electrocardiogram Qt Prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 12 | 15
Gamma-Glutamyltransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 14
Haemoglobin Decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Lipase Increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 35 | 38
Protein Total Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Transaminases Increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 10 | 14
Weight Decreased (Investigations) | 0 | 0 | 1 | 0 | 5 | 1 | 1 | 3 | 51 | 62
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 3 | 4 | 3 | 99 | 111
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 17 | 18
Electrolyte Imbalance (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 4
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 23 | 24
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 6 | 7
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 8 | 10
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 14 | 15
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 11 | 12
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 2 | 1 | 2 | 1 | 34 | 41
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 25 | 30
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 19 | 23
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 19 | 23
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 2 | 31 | 38
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 3 | 1 | 4 | 1 | 56 | 67
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 8 | 9
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 3
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 14 | 15
Fracture Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle Atrophy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 24 | 27
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 17 | 19
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 32 | 33
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 5 | 6
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 2 | 2 | 1 | 1 | 40 | 48
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 12 | 16
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 17
Osteonecrosis Of Jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 1 | 23 | 29
Melanocytic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Akathisia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Complex Partial Seizures (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 38 | 42
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 19 | 23
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 2 | 0 | 3 | 1 | 66 | 74
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 9 | 10
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 5
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Neuropathy Peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 7 | 8
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 23 | 26
Peripheral Motor Neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 4
Sensory Loss (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Sinus Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 20
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 24 | 25
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 16 | 17
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 1 | 45 | 52
Mood Altered (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 6 | 7
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 4
Renal Failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Urinary Incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 5 | 6
Breast Oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Retracted Nipple (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Vaginal Odour (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 3 | 3 | 3 | 0 | 83 | 94
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 14 | 16
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1 | 2 | 5 | 0 | 0 | 61 | 72
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 16 | 18
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 11 | 13
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 4
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 5 | 6
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 2 | 17 | 23
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 33 | 36
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 18 | 18
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 5 | 6
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 13 | 14
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 10 | 11
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 18 | 20
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 5 | 6
Pigmentation Disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 19 | 22
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 39 | 44
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 4
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 3
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Haemodynamic Instability (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hot Flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 5 | 6
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 12 | 14
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 8 | 10
Jugular Vein Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.